CLINICAL TRIAL: NCT03360929
Title: A Phase I/II, Open-label, Multi-center Study to Evaluate Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of AZD3759 in Chinese Patients With EGFRm+ NSCLC With Central Nervous System (CNS) Metastases
Brief Title: Evaluate Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of AZD3759
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LYZZ Alpha Holding Ltd (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZD3759-001
Record Dates: First submitted 2017-11-16; First posted 2017-12-04 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — AZD3759

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open-label, dose escalation and phase II study, consisting of dose escalation study in Part A and phase II study in Part B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental): Study drug: AZD3759 Strength: 50mg/tablet, 100mg/tablet Dose escalation:A treatment cycle consists of consecutive 21 days of dosing. two dose cohorts are planned for dose escalation, including: 150 and 250 mg twice daily.
  RP2D in dose expansion.
  Interventions: Drug: AZD3759

INTERVENTIONS:
Drug: AZD3759 — Strength: 50mg/tablet, 100mg/tablet Dosage and administration: Twice daily administration under fasting state.

SUMMARY:
This is a multi-center, open-label, dose escalation and phase I/II study, consisting of dose escalation in Part A and phase II study in Part B.

DETAILED DESCRIPTION:
Dose escalation and dose expansion to determine safety and tolerability of AZD3759, and explore RP2D in treatment of Chinese patients with EGFRm+ NSCLC with CNS metastasis. Two dose cohorts include: 150 and 250mg twice daily. Subjects will receive multiple doses of AZD3759 for consecutively 21 days each cycle. Dose escalation is planned to be performed in a single center, and dose expansion in multiple centers.

ELIGIBILITY:
Inclusion criteria:

1. Subjects must provide written informed consent before any study related procedure.
2. Male or female Chinese patients ≥18 years old.
3. Histologically or cytologically confirmed non-small cell lung cancer with activating mutation in EGFR gene (including Exon19Del and/or L858R). A validated and robust test method reviewed and approved by the regulatory authority should be used to determine EGFR mutation status in tissue or plasma locally.
4. Patients with advanced non-small cell lung cancer (stage IV) with documented BM and/or LM. Part A dose escalation can include EGFR TKI-naïve NSCLC patients with measurable lung lesion and no BM. Patients with BM and/or LM in each dose group shall account for at least one-third.
5. According to Eastern Cooperative Oncology Group (ECOG) Scale, performance status is grade 0 to 1, without worsening in the past 2 weeks, and life expectancy of at least 3 months. If ECOG performance status is grade 2 due to LM disease, the patient can also be enrolled.
6. Non-surgical sterilized women of child-bearing potential and male subjects shall agree to take medically acceptable contraception measures during dosing of investigational drug and 3 months after completion of study treatment. Non-surgical sterilized women of child-bearing potential must have negative blood pregnancy test at screening.
7. Asymptomatic BM patients who have not received prior treatment with any EGFR TKI or symptomatic BM patients who are not warranted temporally for definitive local treatment (surgery or radiotherapy). For patients with prior local treatment for BM lesion (surgery or radiotherapy), intracranial lesion progression is required.
8. BM patients must have at least one measurable intracranial lesion; in case of prior radiotherapy for BM lesion, progression is required and must meet measurable lesion criteria again. Measurable extracranial disease is not required.
9. LM patients must be confirmed by the presence of malignant cells by cerebrospinal fluid (CSF) cytology. Diagnosis of LM disease by MRI alone does not meet inclusion criteria. Patients with both BM and LM are considered as LM.
10. LM patients must have at least one leptomeningeal lesion which shows visible abnormality by MRI. Measurable extracranial disease is not required.

Exclusion criteria:

Patients meeting any of the following criteria cannot participate in the study:

1. Have taken any other investigational drug in a clinical trial within 30 days prior to initial dose.
2. Prior treatment with any EGFR TKI within 8 days or 5 half-lives of the drug (see table 19 Washout of EGFR TKIs) prior to initial dose of study drug. If the washout period for the EGFR TKI cannot be reached due to schedule or pharmacokinetic properties, an alternative washout period can be proposed based on recovery period of known adverse drug reactions, which must be agreed to in advance by the Investigator and the Sponsor.
3. T790M mutation positive patients.
4. Have received previous treatment regimen including any cytotoxic chemotherapy or other anti-cancer drugs (other than EGFR TKIs) for treatment of advanced non-small cell lung cancer within 14 days prior to initial dose of study drug.
5. Patients with medically uncontrollable seizures and/or untreated (eg., requiring mannitol and/or placement a VP shunt) intracranial hypertension are excluded.
6. Have undergone major surgical procedure (excluding placement of vascular indwelling needle) or serious trauma within 4 weeks prior to initial dose of study drug, or major surgical procedure is expected during the study.
7. Patients who have received radiotherapy for a large area within 4 weeks, or local palliative radiotherapy for a small area within 1 week prior to initial dose of study drug (for subjects requiring radiotherapy for more than 30% bone marrow, the radiotherapy must be completed before 4 weeks prior to initial dose).
8. BM and LM patients who have received whole-brain radiotherapy.
9. Patients with a history of allergy to AZD3759 and its structural analogues (Gefitinib) or pharmaceutical excipients (whether active or not).
10. Subjects who are receiving (or cannot discontinue at least 1 week prior to initial dose of study drug) any drug or traditional Chinese medicine known to inhibit or induce CYP3A4 or CYP3A5 activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 21 days after the first dose
  AE.SAE,vital signs, physical examination,laboratory examinations etc.
anti-tumor activity | every 6 weeks
  ORR, DCR, DOR, PFS and tumor size changing compared with baseline according to RECIST 1.1

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Pre-dose and 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h(C0D2) and 48h(C0D3) after the first single-dose(C0D1) ;Pre-dose of C1D1,C1D8, C1D15, C1D21 and C2D1 and 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h post dose on C1D21 during multiple dosing.
  Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC) | Pre-dose and 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h(C0D2) and 48h(C0D3) after the first single-dose(C0D1) ;Pre-dose of C1D1,C1D8, C1D15, C1D21 and C2D1 and 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h post dose on C1D21 during multiple dosing.
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, Professor, Principal Investigator — Guangdong Provincial People's Hospital
Locations (4):
- China (4):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - 0004, Wuhan, Hubei
  - 0002, Changsha, Hunan
  - 0003, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Taphoorn MJ, Claassens L, Aaronson NK, Coens C, Mauer M, Osoba D, Stupp R, Mirimanoff RO, van den Bent MJ, Bottomley A; EORTC Quality of Life Group, and Brain Cancer, NCIC and Radiotherapy Groups. An international validation study of the EORTC brain cancer module (EORTC QLQ-BN20) for assessing health-related quality of life and symptoms in brain cancer patients. Eur J Cancer. 2010 Apr;46(6):1033-40. doi: 10.1016/j.ejca.2010.01.012. Epub 2010 Feb 22. PMID 20181476
- [Derived] Li K, Chen B, Wang J, Wu L. Long-term survival of a patient with epidermal growth factor receptor (EGFR)-mutant non-small cell lung cancer (NSCLC) and untreated multiple brain metastases treated with zorifertinib: A case report. Thorac Cancer. 2024 Jun;15(16):1325-1329. doi: 10.1111/1759-7714.15317. Epub 2024 Apr 26. PMID 38666433